CLINICAL TRIAL: NCT04736498
Title: Inferior Venacava Ultrasound to Guide Fluid Management for Prevention of Hypotension After Spinal Anesthesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University, Nepal (Other)
Collaborators: Tribhuvan University (Unknown)
Responsible Party: Principal Investigator, Semanta Dahal, MBBS, MD, Tribhuvan University, Nepal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 308/075/076
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Hypotension; Fluid Overload
Keywords: Collapsibility index; Inferior venacava ultrasound; Spinal anesthesia; Transthoracic echocardiography
MeSH Terms: conditions — Hypotension; Edema

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Control group will follow the standard procedure in our centre and will not undergo USG assessment before spinal anaesthesia. The spinal anaesthesia procedure will be standardized. Under strict aseptic precautions spinal anesthesia will be performed at L3-L4 inter-space using a 25 Gauge Quincke spinal needle (B. Braun Medical SA, Melsungen, Germany) in sitting position. 3 ml of hyperbaric bupivacaine 0.5% (15 mg) will be injected with the needle orifice oriented cranially. After injection, patients will be immediately positioned supine. Meanwhile, the non-invasive blood pressure will be measured and recorded every 3 minute for 30 min and then every 5 min throughout surgery and anesthesia.
- USG arm (Experimental): In the IVC USG group, USG assessment and volume optimisation using collapsibility index will be done prior to spinal anaesthesia. all patients will be lying supine, for at least 5 min before IVC examination. Ultrasound measurements will be performed using a Sonosite M-Turbo (Sonosite Inc., USA) machine and phased array 5-1 Megahertz transducer (Sonosite Inc.) set to abdominal mode by an M-mode modality through the subcostal view. All IVC measurements will be performed by principal investigator before spinal anaesthesia. Principal investigator should have performed more than 25 scans before the commencement of the study.
  Interventions: Other: Inferior venacava Ultrasonography (IVC USG) guided fluid management

INTERVENTIONS:
Other: Inferior venacava Ultrasonography (IVC USG) guided fluid management — The IVC will be visualized using a paramedian long-axis view via a subcostal approach. A two-dimensional image of the IVC as it enters the right atrium will be first obtained. Variations in IVC diameter with respiration will be assessed using M-mode imaging performed 2 to 3 cm distal to the junction of right atrium and IVC. Maximum and minimum diameter will be measured from inner wall to inner wall and collapsibility index(CI) will be calculated using formula: CI = [(dIVCmax - dIVCmin)/dIVCmax] x 100% CI of ˃36% will be accepted as predicted fluid responder and ≤36% will be regarded as predicted fluid non responders. Predicted fluid responders will receive a bolus of 500 ml of Ringer's lactate over a time period of 15 min, after which the IVC diameter variation will be reassessed. Additional 250ml of Ringer's lactate bolus will be applied until a non fluid responder pattern is observed during IVC USG. Thereafter,spinal anaesthesia will be performed.
  Arms: USG arm

SUMMARY:
Hypotension is common during spinal anesthesia and contributes to underperfusion and ischemia. Severe episodes of intraoperative hypotension is an independent risk factor for myocardial infarction, stroke, heart failure, acute kidney injury, prolonged hospital stay and increased one year mortality rates. Empiric fluid preloading can be done to decrease the incidence of hypotension but carries risk of fluid overload especially in elderly and cardiac patients. Inferior venacava ultrasonography (IVC USG) has been used in spontaneously breathing critically ill patients for volume responsiveness but there is limited data regarding its use for volume optimization in perioperative setting. The aim of this study is to evaluate the use of inferior venacava ultrasound to guide fluid management for prevention of hypotension after spinal anesthesia.

DETAILED DESCRIPTION:
Introduction:

Hypotension is common during spinal anesthesia and contributes to underperfusion and ischemia. It occurs due to reduction in both cardiac output and systemic vascular resistance. Even short duration of intraoperative MAP less than 55 mmHg has been found to be associated with Acute kidney injury (AKI) and myocardial injury. Severe episodes of intraoperative hypotension is an independent risk factor for myocardial infarction, stroke, heart failure, acute kidney injury, prolonged hospital stay and increased 1 year mortality rates. Predictive variables for spinal anesthesia induced hypotension includes peak sensory level, chronic alcohol consumption, emergency surgery, age more than 40 years, hypertension, combined spinal/general anaesthesia(GA), spinal puncture at or above lumbar 2 lumber 3 (L2L3) interspace. Preoperative volume status is an important factor determining patient's hemodynamic status. Traditional static parameters such as central venous pressure have been criticized for invasiveness and lack of accuracy. Newer noninvasive dynamic parameters like inferior venacava diameter and Collapsibility index(CI), acoustic echocardiography, stroke volume variation and pulse pressure variation etc are being used widely for assessing volume status.

Study Objective: To evaluate the use of inferior vena cava ultrasound to guide fluid management for prevention of hypotension after spinal anesthesia.

Design: A randomized prospective interventional study

Sample size: 92

Place: Operating theatres of Tribhuvan University Teaching Hospital (TUTH), Maharajgunj Medical Campus (MMC), Institute of Medicine (IOM).

Interventions: A total of 92 patients undergoing lower limb orthopedic surgery will be enrolled in the study. They will be randomized into USG group and Control group. In the USG group, IVC ultrasound will be done and collapsibility index (CI) will be calculated. Depending upon the value of calculated CI, fluid management will be done by infusing Ringer's Lactate (RL). Thereafter spinal anesthesia will be performed. In the control group, spinal anesthesia will be performed without IVC USG assessment. In both the groups, incidence of hypotension and amount of fluid and vasopressors administered will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥16-65 years
2. American Society of Anaesthesiology physical status (ASA PS) I and II
3. Requiring elective spinal anaesthesia for lower limb orthopaedic surgery

Exclusion Criteria:

1. Patients with pre-procedural hypotension, defined as two consecutive measurements of systolic arterial pressure (SAP) less than 90 mmHg or mean arterial pressure (MAP) less of 60 mmHg.
2. Contraindication for Spinal Anaesthesia

   * Platelet counts ˂100,000 per microlitre of blood
   * International normalized ratio (INR) ≥1.5
   * Bleeding disorders
   * Infection at injection site

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Comparison of incidence of hypotension between two groups | 30 minutes after spinal anaesthesia
  To compare the incidence of hypotension after spinal anesthesia between two groups, USG group who have undergone volemic optimization after USG assessment and control group.

SECONDARY OUTCOMES:
Analyse amount of fluids administered between two groups | 30 minutes after spinal anaesthesia
  To compare fluid adjustment requirement between USG group and control group
Compare vasopressors used between two groups | 30 minutes after spinal anaesthesia
  To compare the rate of vasopressors used between USG group and control group

CONTACTS AND LOCATIONS:
Overall Officials: Semanta Dahal, MBBS, MD, Principal Investigator — Institute of Medicine (IOM), Tribhuvan University
Locations (1):
- Semanta Dahal, Maharajgunj, Bagmati, Nepal

REFERENCES:
- [Background] Wulf HF. The centennial of spinal anesthesia. Anesthesiology. 1998 Aug;89(2):500-6. doi: 10.1097/00000542-199808000-00028. No abstract available. PMID 9710410
- [Background] Brull R, Macfarlane A, Chan V. Spinal, epidural and caudal anesthesia. In: Miller RD, editor. Miller's anesthesia. 8th ed: Elsevier; 2015.
- [Background] Carpenter RL, Caplan RA, Brown DL, Stephenson C, Wu R. Incidence and risk factors for side effects of spinal anesthesia. Anesthesiology. 1992 Jun;76(6):906-16. doi: 10.1097/00000542-199206000-00006. PMID 1599111
- [Background] Salinas FV, Sueda LA, Liu SS. Physiology of spinal anaesthesia and practical suggestions for successful spinal anaesthesia. Best Pract Res Clin Anaesthesiol. 2003 Sep;17(3):289-303. doi: 10.1016/s1521-6896(02)00114-3. PMID 14529003
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Sun LY, Wijeysundera DN, Tait GA, Beattie WS. Association of intraoperative hypotension with acute kidney injury after elective noncardiac surgery. Anesthesiology. 2015 Sep;123(3):515-23. doi: 10.1097/ALN.0000000000000765. PMID 26181335
- [Background] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Background] Zhang J, Critchley LA. Inferior Vena Cava Ultrasonography before General Anesthesia Can Predict Hypotension after Induction. Anesthesiology. 2016 Mar;124(3):580-9. doi: 10.1097/ALN.0000000000001002. PMID 26771910
- [Background] Monk TG, Bronsert MR, Henderson WG, Mangione MP, Sum-Ping ST, Bentt DR, Nguyen JD, Richman JS, Meguid RA, Hammermeister KE. Association between Intraoperative Hypotension and Hypertension and 30-day Postoperative Mortality in Noncardiac Surgery. Anesthesiology. 2015 Aug;123(2):307-19. doi: 10.1097/ALN.0000000000000756. PMID 26083768
- [Background] Chappell D, Jacob M, Hofmann-Kiefer K, Conzen P, Rehm M. A rational approach to perioperative fluid management. Anesthesiology. 2008 Oct;109(4):723-40. doi: 10.1097/ALN.0b013e3181863117. PMID 18813052
- [Background] Bajwa SJ, Kulshrestha A, Jindal R. Co-loading or pre-loading for prevention of hypotension after spinal anaesthesia! a therapeutic dilemma. Anesth Essays Res. 2013 May-Aug;7(2):155-9. doi: 10.4103/0259-1162.118943. PMID 25885825
- [Background] Minto G, Scott MJ, Miller TE. Monitoring needs and goal-directed fluid therapy within an enhanced recovery program. Anesthesiol Clin. 2015 Mar;33(1):35-49. doi: 10.1016/j.anclin.2014.11.003. PMID 25701927
- [Background] Doherty M, Buggy DJ. Intraoperative fluids: how much is too much? Br J Anaesth. 2012 Jul;109(1):69-79. doi: 10.1093/bja/aes171. Epub 2012 Jun 1. PMID 22661747
- [Background] Singh J, Ranjit S, Shrestha S, Sharma R, Marahatta SB. Effect of preloading on hemodynamic of the patient undergoing surgery under spinal anaesthesia. Kathmandu Univ Med J (KUMJ). 2010 Apr-Jun;8(30):216-21. doi: 10.3126/kumj.v8i2.3562. PMID 21209539
- [Background] Marik PE, Baram M, Vahid B. Does central venous pressure predict fluid responsiveness? A systematic review of the literature and the tale of seven mares. Chest. 2008 Jul;134(1):172-8. doi: 10.1378/chest.07-2331. PMID 18628220
- [Background] Kalantari K, Chang JN, Ronco C, Rosner MH. Assessment of intravascular volume status and volume responsiveness in critically ill patients. Kidney Int. 2013 Jun;83(6):1017-28. doi: 10.1038/ki.2012.424. Epub 2013 Jan 9. PMID 23302716
- [Background] Lansdorp B, Lemson J, van Putten MJ, de Keijzer A, van der Hoeven JG, Pickkers P. Dynamic indices do not predict volume responsiveness in routine clinical practice. Br J Anaesth. 2012 Mar;108(3):395-401. doi: 10.1093/bja/aer411. Epub 2011 Dec 20. PMID 22185905
- [Background] Muller L, Bobbia X, Toumi M, Louart G, Molinari N, Ragonnet B, Quintard H, Leone M, Zoric L, Lefrant JY; AzuRea group. Respiratory variations of inferior vena cava diameter to predict fluid responsiveness in spontaneously breathing patients with acute circulatory failure: need for a cautious use. Crit Care. 2012 Oct 8;16(5):R188. doi: 10.1186/cc11672. PMID 23043910
- [Background] Lamia B, Ochagavia A, Monnet X, Chemla D, Richard C, Teboul JL. Echocardiographic prediction of volume responsiveness in critically ill patients with spontaneously breathing activity. Intensive Care Med. 2007 Jul;33(7):1125-1132. doi: 10.1007/s00134-007-0646-7. Epub 2007 May 17. PMID 17508199
- [Background] Corl KA, George NR, Romanoff J, Levinson AT, Chheng DB, Merchant RC, Levy MM, Napoli AM. Inferior vena cava collapsibility detects fluid responsiveness among spontaneously breathing critically-ill patients. J Crit Care. 2017 Oct;41:130-137. doi: 10.1016/j.jcrc.2017.05.008. Epub 2017 May 12. PMID 28525778
- [Background] Zhang Z, Xu X, Ye S, Xu L. Ultrasonographic measurement of the respiratory variation in the inferior vena cava diameter is predictive of fluid responsiveness in critically ill patients: systematic review and meta-analysis. Ultrasound Med Biol. 2014 May;40(5):845-53. doi: 10.1016/j.ultrasmedbio.2013.12.010. Epub 2014 Feb 2. PMID 24495437
- [Background] Preau S, Bortolotti P, Colling D, Dewavrin F, Colas V, Voisin B, Onimus T, Drumez E, Durocher A, Redheuil A, Saulnier F. Diagnostic Accuracy of the Inferior Vena Cava Collapsibility to Predict Fluid Responsiveness in Spontaneously Breathing Patients With Sepsis and Acute Circulatory Failure. Crit Care Med. 2017 Mar;45(3):e290-e297. doi: 10.1097/CCM.0000000000002090. PMID 27749318
- [Background] Di Pietro S, Falaschi F, Bruno A, Perrone T, Musella V, Perlini S. The learning curve of sonographic inferior vena cava evaluation by novice medical students: the Pavia experience. J Ultrasound. 2018 Jun;21(2):137-144. doi: 10.1007/s40477-018-0292-7. Epub 2018 Mar 21. PMID 29564661
- [Background] Szabo M, Bozo A, Darvas K, Horvath A, Ivanyi ZD. Role of inferior vena cava collapsibility index in the prediction of hypotension associated with general anesthesia: an observational study. BMC Anesthesiol. 2019 Aug 7;19(1):139. doi: 10.1186/s12871-019-0809-4. PMID 31390983
- [Background] Ceruti S, Anselmi L, Minotti B, Franceschini D, Aguirre J, Borgeat A, Saporito A. Prevention of arterial hypotension after spinal anaesthesia using vena cava ultrasound to guide fluid management. Br J Anaesth. 2018 Jan;120(1):101-108. doi: 10.1016/j.bja.2017.08.001. Epub 2017 Nov 23. PMID 29397116
- [Background] Salama ER, Elkashlan M. Pre-operative ultrasonographic evaluation of inferior vena cava collapsibility index and caval aorta index as new predictors for hypotension after induction of spinal anaesthesia: A prospective observational study. Eur J Anaesthesiol. 2019 Apr;36(4):297-302. doi: 10.1097/EJA.0000000000000956. PMID 30664523
- [Background] Chinachoti T, Tritrakarn T. Prospective study of hypotension and bradycardia during spinal anesthesia with bupivacaine: incidence and risk factors, part two. J Med Assoc Thai. 2007 Mar;90(3):492-501. PMID 17427526